CLINICAL TRIAL: NCT06183242
Title: Multicenter Comparative Randomized Study to Assess Safety and Efficacy and Select the Optimal Dosage Regimen of REMAXA®, Enteric-coated Tablets, in Comparison With REMAXOL®, Solution for Infusions, in Patients With Intrahepatic Cholestasis Caused by Chronic Diffuse Liver Diseases
Brief Title: Comparative Study of REMAXA®, Enteric-coated Tablets and REMAXOL®, Solution for Infusions, in Intrahepatic Cholestasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RXA-II-III-Chol-2022
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-01

CONDITIONS: Cholestasis, Intrahepatic
Keywords: intrahepatic cholestasis; chronic diffuse liver disease; Biliary Stasis, Intrahepatic
MeSH Terms: conditions — Cholestasis, Intrahepatic | interventions — Inosine; Methionine; Niacinamide; Succinic Acid; Remaxol; Meglumine

STUDY DESIGN:
Intervention Model Description: Multicenter prospective two-stage comparative randomized parallel group study with placebo control
Who Masked: Participant, Care Provider
Masking Description: On stage 1, there will be no blinding (because REMAXOL is a solution for infusions). On stage 2, blinding will be ensured by placebo masking and drug assignment via IWRS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group I-1 (Experimental): Intake of REMAXA, enteric-coated tablets, 2 tablets 3 times a day for 10 days
  Interventions: Drug: Remaxa, enteric-coated tablets
- Group I-2 (Experimental): Intake of REMAXA, enteric-coated tablets, 2 tablets 2 times a day for 10 days
  Interventions: Drug: Remaxa, enteric-coated tablets
- Group I-3 (Experimental): Intake of REMAXA, enteric-coated tablets, 2 tablets once a day for 10 days
  Interventions: Drug: Remaxa, enteric-coated tablets
- Group I-4 (Active Comparator): Infusions of REMAXOL, solution for infusion, by intravenous drip, 400 ml once a day for 10 days.
  Interventions: Drug: Remaxol
- Group II-1 (Experimental): Intake of REMAXA, enteric-coated tablets, during 10 days according to optimal dosing regimen established during stage I.
  Interventions: Drug: Remaxa, enteric-coated tablets
- Group II-2 (Active Comparator): Infusions of REMAXOL, solution for infusion, by intravenous drip, 400 ml once a day for 10 days.
  Interventions: Drug: Remaxol
- Group II-3 (Placebo Comparator): Intake of Placebo, enteric-coated tablets, during 10 days, analogous to dosing regimen in Group II-1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remaxa, enteric-coated tablets — enteric-coated tablets
  Other Names: inosine, methionine, nicotinamide, succinic acid
  Arms: Group I-1; Group I-2; Group I-3; Group II-1
Drug: Remaxol — solution for infusions
  Other Names: inosine + meglumine + methionine + nicotinamide + succinic acid
  Arms: Group I-4; Group II-2
Drug: Placebo — enteric-coated tablets
  Arms: Group II-3

SUMMARY:
Chronic diffuse liver disease implies liver damage of various origin - viral hepatitis, the effect of xenobiotics (alcohol, drugs, medications, industrial toxins), metabolic disorders, non-alcoholic fatty liver disease. Intrahepatic cholestasis syndrome, or bile retention, occurs in 11-55% of cases of diffuse chronic liver diseases, usually leads to a worsening of the liver disease, a decrease in the effectiveness of treatment. The drug REMAXOL® is a solution for infusion, which has shown high effectiveness in the syndrome of intrahepatic cholestasis in cases of liver dysfunction due to acute or chronic damage. The study drug REMAXA® enteric-coated tablets is a hybrid drug which contains the same active metabolites as REMAXOL, i.e. inosine, methionine, nicotinamide, and succinic acid. The purpose of this study is to select the optimal dose and dosage regimen followed by evaluation safety and efficacy of REMAXA®, enteric-coated tablets, in comparison with REMAXOL®, solution for infusion, in patients who suffer from chronic diffuse liver diseases and have intrahepatic cholestasis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 70 years (inclusive).
2. Patients with intrahepatic cholestasis syndrome in chronic diffuse liver diseases (alcoholic liver disease, toxic damage liver, liver fibrosis and sclerosis, fatty liver degeneration, chronic hepatitis) and/or with other liver dysfunction due to acute or chronic damage (toxic, alcoholic, viral, drug hepatitis).
3. Gamma-glutamyl transpeptidase (GGTP) exceeds the upper normal limit by 3 times or more and/or alkaline phosphatase (ALP) exceeds the upper normal limit by 1.5 times or more.
4. Negative pregnancy test in female patients.
5. Consent to the use of adequate contraceptive methods or complete abstinence from sexual activity for the study period.
6. Agreement to limit alcohol consumption to a maximum of 2 units alcohol per month (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of dry wine or 50 ml strong alcoholic drinks), or complete abstinence from drinking alcohol for period of the study.
7. Signed informed consent.

Exclusion Criteria:

1. Cirrhotic stage of chronic liver disease (Class A-C by Child-Pugh).
2. Hyperbilirubinemia more than 100 µmol/l.
3. GGTP level is more than 10 upper normal limits.
4. History of autoimmune liver disease.
5. Acute viral hepatitis (B, C, D).
6. Any somatic diseases in the stage of decompensation.
7. Regular use by the patient of medications prohibited in within the framework of this study, within 4 weeks before inclusion in the study and at throughout this study.
8. Hypersensitivity and/or intolerance to any component of the study drug /comparator drug.
9. Pregnancy or lactation period.
10. Peptic ulcer of the stomach and/or duodenum, and/or erosive gastritis in the acute phase.
11. History of chronic kidney disease C4-C5 and/or known glomerular filtration rate <30 ml/min.
12. Regular intake of more than 2 units. alcohol per week.
13. Unstable angina.
14. Myocardial infarction 3 months or less before the expected date of inclusion.
15. Chronic heart failure of III-IV functional class by New York Heart Association (NYHA) classification.
16. History of cancer within the last 5 years, mental illness, HIV infection, tuberculosis, drug addiction.
17. Mental, physical and other reasons that prevent the patient adequately behave and correctly fulfill the conditions of the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Proportion of responders to treatment in the study groups | 11 days
  The proportion of patients who responded to therapy, as indicated by any of the changes of laboratory parameters: a decrease in the level of gamma-glutamyltranspeptidase by at least 40% from the initial level and/or a decrease in the level of alkaline phosphatase by at least 30% from the initial level and/or a decrease in the level of total bilirubin not by less than 30% from the initial to the end of the therapeutic course in the REMAXA group compared to REMAXOL group.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana V Kharitonova, MD PhD, Study Director — STPF POLYSAN
Locations (3):
- Russia (3):
  - Research Center for Eco-safety, Ltd., Saint Petersburg
  - City Hospital of the Holy Martyr Elizabeth, Saint Petersburg
  - Medical Company "Hepatologist" Ltd., Samara

IPD SHARING:
Plan to Share IPD: No